CLINICAL TRIAL: NCT03036202
Title: Pharmacokinetic Study of Epinephrine During Cardiac Arrest Determining T1/2 and Time to Peak Concentration
Brief Title: Pharmacokinetics of Epinephrine During Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1471-74
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest
Keywords: epinephrine
MeSH Terms: conditions — Heart Arrest | interventions — Epinephrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples with determination of medical concentration in plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- one group: All patients treated for cardiac arrest, meeting our inclusions criteria will be enrolled in the study. No interventions regarding the national guidelines will be jeopardized, as the plasma concentration following a single dose of epinephrine will be measured in all patient.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — This is truly an observational study to determine T1/2 for epinephrine and time to peak concentration following a single dose of epinephrine in a cardiac arrest setting
  Other Names: Adrenaline

SUMMARY:
To determine the pharmacokinetics of epinephrine during cardiac arrest.

DETAILED DESCRIPTION:
The aim of out study is to determine the pharmacokinetics in humans during cardiac arrest, following a single dose of epinephrine. Venous samples will be withdrawn every minute the first five minutes following a single dose.

The aim of the study is to determine T1/2 in a clinical setting and to determine time to peak concentration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 yrs
* Witnessed non-traumatic cardiac arrest.
* Probable cardiac origin
* Treated by Bergen Emergency Medical Services

Exclusion Criteria:

* Terminal illness
* Residents of nursery homes
* Obvious dead
* Hypothermic patients
* Epinephrine administered before arrival of study physician

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac arrest of an assumed cardiac origin, treated by the Bergen Emergency Medical Service.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Concentration of epinephrine (ng/mL) as a function of time the first five minutes following administration | Blood samples will be drawn within minutes, and the survivors transported to hospital. The data according to Utstein-style, will also be collected. Blood samples will be analysed within weeks.Total timeframe for the study is estimated to one year.
  Blood concentration of epinephrine will be determined the first five minutes following administration. For every minute starting With administration of epinephrine, blood samples will be drawn to determine the concentration (ng/mL). In total, six samples will be drawn. The administered dose (1 mg) will also be related to the patients weight, either estimated, or for those survivors admitted to hospital, measured in the Intensive Care Unit. Further, data according to the Utstein-template will be recorded.However, the primary outcome is to determine the plasma concentrations in every patients the first five minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Baard E Heradstveit, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, N, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available to other researchers. The data will be presented pooled and anonymously